CLINICAL TRIAL: NCT02631720
Title: A Prospective Multicenter Observational Cohort Study to Define the Risks Factors, Mechanisms, and Manifestations of Chronic Lung Allograft Dysfunction (CLAD) Phenotypes (CTOT-20)
Brief Title: CLAD Phenotype Specific Risk Factors and Mechanisms
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOT-20
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Lung Transplant; Post Lung Transplantation
Keywords: Chronic Lung Allograft Dysfunction (CLAD); Restrictive chronic lung allograft dysfunction (RCLAD); Bronchiolitis Obliterans Syndrome (BOS); CLAD risk factors; observational study
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Blood Specimen Collection; Phlebotomy; Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral whole blood samples: DNA, RNA, Plasma, Serum Bronchoalveolar lavage (BAL): aliquots with DNA, cells, supernatant
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adult Lung Transplant Recipients: Adult lung transplant recipients undergoing lung transplant at each of the participating centers.
  Interventions: Procedure: Blood Draw; Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Blood Draw
  Other Names: Phlebotomy; Venipuncture
Procedure: Bronchoscopy

SUMMARY:
While many patients experience benefits from transplant, complications such as infections and lung rejection may affect long term survival and quality of life. In this study doctors are looking at a complication called Chronic Lung Allograft Dysfunction (CLAD). CLAD is thought to be chronic rejection of the lung by the immune system and is the leading cause of death after lung transplantation.

The purpose of this study is to help doctors determine:

* why some people get CLAD and others do not
* how patients who get CLAD do after CLAD is diagnosed
* how CLAD may affect quality of life

DETAILED DESCRIPTION:
This is an observational, prospective, multicenter study of newly transplanted adult, first lung transplant recipients that will collect longitudinal clinical data, patient reported quality of life (QOL) data, and serial biological samples to determine the risk factors, pathophysiology, and manifestations of restrictive chronic lung allograft dysfunction (RCLAD) and bronchiolitis obliterans syndrome (BOS). Anticipated participant accrual is within three years of study start-up. The total study duration is four years. Participants will be followed a minimum of 1 and a maximum of 4 years.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as study participants:

1. Subject must be able to understand and provide written informed consent and

   -Must be ≥18 years of age at the time of written informed consent.
2. Anticipated listing for lung transplantation OR within 45 days of having received a single or bilateral cadaveric donor lung transplant.

   - Enrollment must occur prior to the start of bronchoscopies eligible for research bronchoalveolar lavage (BAL) sampling.
3. Undergoing first lung transplant operation.
4. Transplant surgery to be performed or performed at enrolling center.

   * Note: Concurrent participation in immune monitoring studies or interventional device trials are permitted.

Exclusion Criteria:

Individuals who meet any of the following criteria are not eligible for enrollment as study participants:

1. Multi-organ recipient.
2. Prior recipients of any solid organ transplant, including prior lung transplant.
3. Prior or concurrent recipient of bone marrow transplant.
4. HIV infection.
5. Any condition which the investigators feel would make it unlikely for the recipient to complete follow up procedures or complete the study.
6. Participation in an investigational drug trial at the time of enrollment visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult lung transplant recipients undergoing lung transplant at each of the participating centers.
Sampling Method: Probability Sample
Enrollment: 884 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Time from transplant to Restrictive Chronic Lung Allograft Dysfunction (RCLAD) or Bronchiolitis Obliterans Syndrome (BOS). | 90 days post-transplant until study completion or participant withdrawal (up to 4 years post-transplant)
  First occurrence of either phenotype.

SECONDARY OUTCOMES:
Longitudinal Quality of life (QOL) trajectory | Baseline until study completion or participant withdrawal (up to 4 years post-transplant)
  As serially assessed by the 36-item Short Form Survey (SF-36) and the St. George's Respiratory Questionnaire (SGRQ)
Mechanistic: Chemokine/cytokine Quantification of Type 1 and Type 17 immune profile proteins | Baseline until study completion or participant withdrawal (up to 4 years post-transplant)
  Measured in the Bronchoalveolar lavage (BAL) supernatant.using standard Luminex and ELISA commercial assays

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Palmer, MD, MHS, Principal Investigator — Duke University; John Belperio, MD, Study Chair — University of California, Los Angeles
Locations (5):
- United States (4):
  - University of California, Los Angeles, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Todd JL, Weigt SS, Neely ML, Grau-Sepulveda MV, Mason K, Sever ML, Kesler K, Kirchner J, Frankel CW, Martinu T, Shino MY, Jackson AM, Pavlisko EN, Williams N, Robien MA, Singer LG, Budev M, Tsuang W, Shah PD, Reynolds JM, Snyder LD, Belperio JA, Palmer SM. Prognosis and Risks for Probable Chronic Lung Allograft Dysfunction: A Prospective Multicenter Study. Am J Respir Crit Care Med. 2025 Feb;211(2):239-247. doi: 10.1164/rccm.202403-0568OC. PMID 39470452
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Clinical Trials in Organ Transplantation (CTOT) — http://www.ctotstudies.org/